CLINICAL TRIAL: NCT02435524
Title: Alive & Thrive Evaluation in Burkina Faso
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: FHI 360 (Other); Centre Muraz (Other); AFRICSanté (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 9066
Record Dates: First submitted 2015-04-22; First posted 2015-05-06 (Estimated); Results first posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2017-08

CONDITIONS: Breast Feeding; Breast Feeding, Exclusive
Keywords: Breast Feeding, Exclusive; Infant Nutrition; Burkina Faso
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A&T Intervention Communes (Experimental)
  Interventions: Behavioral: A&T infant and young child feeding intervention
- Control Communes (No Intervention)

INTERVENTIONS:
Behavioral: A&T infant and young child feeding intervention — 1. Interpersonal communication delivered by community workers and volunteers during home visits and at monthly mother's group meetings to:
     * Increase mother's knowledge about optimal breastfeeding and its benefits
     * Increase mother's self-efficacy related to breastfeeding
     * Improve mother's perceptions about social norms relating to breastfeeding
  2. Community mobilisation activities to:
     - Raise awareness of the benefits of optimal breastfeeding among opinion leaders, and family members, and increase the support they provide to breastfeeding mothers
  3. Enhanced training of government health workers in infant and young child feeding to:
     * Improve their ability to support mothers and provide timely information about infant feeding
  Arms: A&T Intervention Communes

SUMMARY:
The time between birth and age 24 months provides a unique opportunity to impact the long-term health and development of children through improved infant and young child feeding practices. In Burkina Faso, the prevalence of exclusive breastfeeding is currently around 25% in infants younger than six months.

The purpose of this study is to evaluate whether the Alive & Thrive intervention package, consisting of interpersonal counselling and community mobilisation activities, can increase the exclusive breastfeeding rate among infants younger than six months to at least 50% using a cluster randomised design.

ELIGIBILITY:
Inclusion Criteria:

* Gives informed consent
* Being aged from 15 to 49 years old (women of reproductive age)
* Has at least one infant less than 12 months old who is currently alive and lives with her.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 4541 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Filippi, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (2):
- Burkina Faso (2):
  - AFRICSanté, Bobo-Dioulasso
  - Centre Muraz Research Institute, Bobo-Dioulasso

REFERENCES:
- [Derived] Cresswell JA, Ganaba R, Sarrassat S, Some H, Diallo AH, Cousens S, Filippi V. The effect of the Alive & Thrive initiative on exclusive breastfeeding in rural Burkina Faso: a repeated cross-sectional cluster randomised controlled trial. Lancet Glob Health. 2019 Mar;7(3):e357-e365. doi: 10.1016/S2214-109X(18)30494-7. PMID 30784636

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Rural communes were randomised in this study. There are 47 communes in Boucle du Mouhoun; 6 urban communes were excluded leaving 41 rural communes to be randomised to either the intervention or control arm. Of these, 2 intervention and 2 control communes were excluded due to co-intervention.
Units Other Than Participants: Communes
Groups:
- A&T Intervention Communes: Communes where the A&T infant and young child feeding intervention was implemented:
  1. Interpersonal communication delivered by community workers and volunteers during home visits and at monthly mother's group meetings to:
     * Increase mother's knowledge about optimal breastfeeding and its benefits
     * Increase mother's self-efficacy related to breastfeeding
     * Improve mother's perceptions about social norms relating to breastfeeding
  2. Community mobilisation activities to:
     - Raise awareness of the benefits of optimal breastfeeding among opinion leaders, and family members, and increase the support they provide to breastfeeding mothers
  3. Enhanced training of government health workers in infant and young child feeding to:
     * Improve their ability to support mothers and provide timely information about infant feeding
- Control Communes: No intervention
Period: Baseline Survey
Arm/Group | A&T Intervention Communes | Control Communes
Started | 1111; 18 Communes | 1177; 19 Communes
Completed | 1111; 18 Communes (Design: 2 independent cross-sectional surveys; baseline & endline participants not same individuals) | 1177; 19 Communes (Design: 2 independent cross-sectional surveys; baseline & endline participants not same individuals)
Not Completed | 0; 0 Communes | 0; 0 Communes
Period: Endline Survey
Arm/Group | A&T Intervention Communes | Control Communes
Started | 1092; 18 Communes | 1161; 19 Communes
Completed | 1092; 18 Communes (Design: 2 independent cross-sectional surveys; baseline & endline participants not same individuals) | 1161; 19 Communes (Design: 2 independent cross-sectional surveys; baseline & endline participants not same individuals)
Not Completed | 0; 0 Communes | 0; 0 Communes

BASELINE CHARACTERISTICS:
Groups:
- A&T Intervention Communes: Baseline; A&T Intervention Communes: Endline: Communes where the A&T infant and young child feeding intervention was implemented:
  1. Interpersonal communication delivered by community workers and volunteers during home visits and at monthly mother's group meetings to:
     * Increase mother's knowledge about optimal breastfeeding and its benefits
     * Increase mother's self-efficacy related to breastfeeding
     * Improve mother's perceptions about social norms relating to breastfeeding
  2. Community mobilisation activities to:
     - Raise awareness of the benefits of optimal breastfeeding among opinion leaders, and family members, and increase the support they provide to breastfeeding mothers
  3. Enhanced training of government health workers in infant and young child feeding to:
     * Improve their ability to support mothers and provide timely information about infant feeding
- Control Communes: Baseline; Control Communes: Endline: No intervention
- Total: Total of all reporting groups
Arm/Group | A&T Intervention Communes: Baseline | Control Communes: Baseline | A&T Intervention Communes: Endline | Control Communes: Endline | Total
Number analyzed (Participants) | 1111 | 1177 | 1092 | 1161 | 4541
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 39 | 49 | 53 | 43 | 184
  Between 18 and 65 years | 1072 | 1128 | 1039 | 1118 | 4357
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1111 | 1177 | 1092 | 1161 | 4541
  Male | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Burkina Faso | 1111 | 1177 | 1092 | 1161 | 4541

OUTCOME MEASURES:

1. Primary Outcome: Exclusive Breastfeeding on the Day Preceding the Interview as Assessed by Cross Sectional Survey
Description: The percentage of infants aged less than 6 months who were exclusively breastfed on the day preceding the interview.
Time Frame: Infants up to 6 months in a cross-sectional endline survey scheduled for April - July 2017
Population: Endline survey participants with infant aged less than 6 months
Measure: Number (95% Confidence Interval); unit: percentage of exclusive breastfeeding
Arm/Group | A&T Intervention Communes | Control Communes
Number analyzed (Participants) | 552 | 584
percentage of exclusive breastfeeding | 0.933 [0.900 to 0.970] | 0.512 [0.421 to 0.603]

2. Secondary Outcome: Breastfeeding Within 1 Hour of Birth as Assessed by Cross Sectional Survey
Description: The proportion of newborns aged less than 6 months who were breastfed within 1 hour of birth.
Time Frame: Infants up to 6 months in a cross-sectional endline survey scheduled for April - July 2017
Reporting Status: Not Posted

3. Secondary Outcome: Colostrum Given as Assessed by Cross Sectional Survey
Description: The proportion of newborns aged less than 6 months who were given colostrum.
Time Frame: Infants up to 6 months in a cross-sectional endline survey scheduled for April - July 2017
Reporting Status: Not Posted

4. Secondary Outcome: Pre-lacteal Feeds as Assessed by Cross Sectional Survey
Description: The proportion of newborns aged less than 6 months who received no pre-lacteal feeds before breastfeeding was established
Time Frame: Infants up to 6 months in a cross-sectional endline survey scheduled for April - July 2017
Reporting Status: Not Posted

5. Secondary Outcome: Semi-solid, Solid or Soft Foods Consumed in the Previous Day as Assessed by Cross Sectional Survey
Description: The proportion of infants age 6 to 8 months who received semi-solid, solid or soft foods in the previous day.
Time Frame: Infants age 6-8 months in a cross-sectional endline survey scheduled for April - July 2017
Reporting Status: Not Posted

6. Secondary Outcome: Minimum Acceptable Diet (Apart From Breast Milk) on the Day Preceding Interview as Assessed by Cross Sectional Survey
Description: The proportion of infants aged 6 to 11.9 months who received a minimum acceptable diet (apart from breast milk) on the day preceding interview.
Time Frame: Infants age 6-11.9 months in a cross-sectional endline survey scheduled for April - July 2017
Reporting Status: Not Posted

7. Secondary Outcome: Dietary Diversity as Assessed by Cross Sectional Survey
Description: Dietary diversity among infants age 6 to 11.9 months.
Time Frame: Infants age 6-11.9 months in a cross-sectional endline survey scheduled for April - July 2017
Reporting Status: Not Posted

8. Secondary Outcome: Breast Milk on the Day Preceding the Interview as Assessed by Cross Sectional Survey
Description: The proportion of children aged 6 to 11.9 months who were fed breast milk on the day preceding the interview.
Time Frame: Infants age 6-11.9 months in a cross-sectional endline survey scheduled for April - July 2017
Reporting Status: Not Posted

9. Secondary Outcome: Mother's Accurate Knowledge of Good Breastfeeding Practice as Assessed by Cross Sectional Survey
Description: Mother's accurate knowledge of:
  * Optimal timing of breastfeeding initiation
  * Optimal duration of exclusive breastfeeding
  * Benefits of optimal breastfeeding practices for the infant
  * Solutions to common difficulties, for example engorgement, cracked and sore nipples
  * Optimal timing to introduce complementary feeding
  * Optimal dietary diversity and frequency of complementary feeding up to 12 months
Time Frame: Mothers of infants aged up to 12 months in a cross-sectional endline survey scheduled for April - July 2017
Reporting Status: Not Posted

10. Secondary Outcome: Mother's Self-reported Breastfeeding Practices as Assessed by Cross Sectional Survey
Description: Mother's self-reported breastfeeding practices, including asking her if she experiences any barriers or difficulties with breastfeeding such as engorgement, cracked and sore nipples, or breastfeeding when working outside of the home.
Time Frame: Mothers of infants aged up to 12 months in a cross-sectional endline survey scheduled for April - July 2017
Reporting Status: Not Posted

11. Secondary Outcome: Mother's Perceptions and Beliefs Surrounding Breastfeeding
Description: Mother's perceptions and beliefs about breastfeeding (qualitative component).
Time Frame: Mothers of infants aged up to 12 months in a cross-sectional endline survey scheduled for April - July 2017
Reporting Status: Not Posted

12. Secondary Outcome: Knowledge, Beliefs and Perceptions Surrounding Breastfeeding of Family Members
Description: Knowledge, beliefs and perceptions of family members, such as mothers or mothers in law, community opinion leaders towards optimal infant and child feeding practices (qualitative component).
Time Frame: Family members of infants aged up to 12 months in a cross-sectional endline survey scheduled for April - July 2017
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Two cross sectional surveys: baseline (2015) & endline (2017)
Arm/Group | A&T Intervention Communes | Control Communes
All-Cause Mortality (participants affected / at risk) | 0/2203 | 0/2338
Serious Adverse Events (participants affected / at risk) | 0/2203 | 0/2338
Other Adverse Events (participants affected / at risk) | 0/2203 | 0/2338

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-16): https://cdn.clinicaltrials.gov/large-docs/24/NCT02435524/Prot_SAP_000.pdf